CLINICAL TRIAL: NCT01654679
Title: Impact of Preoperative Local Water-Filtered Infrared-A (wIRA) Irradiation on Postoperative Wound Healing - A Randomized Patient- and Observer Blinded Controlled Clinical Trial
Brief Title: Impact of Preoperative Local Water-Filtered Infrared-A (wIRA) Irradiation on Postoperative Wound Healing
Acronym: Hydrosun
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Research Foundation (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Mark Hartel, Priv.-Doz. Dr. med., German Research Foundation
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: HydrosunWoundHealing
Record Dates: First submitted 2012-07-22; First posted 2012-08-01 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Wound Infection Rate After Surgery; Impact of Wound Infection on Pain and Wound Healing
Keywords: wound infection; surgery; surgical wound infection rate; wound healing
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- wIRA irradiation (Active Comparator): Patients in Group A received local water-filtered infrared A (wIRA) irradiation once for 20 min preoperatively.
  Interventions: Device: wIRA irradiation
- visible light only (Sham Comparator): Patients assigned to Group B only received normal visible light application for 20 min prior to surgery.
  Interventions: Other: visible light only

INTERVENTIONS:
Device: wIRA irradiation — wIRA irradiation for 20min prior to surgery. The distance between the light bulb and the skin surface was 27cm.
  Other Names: wIRA (Hydrosun® radiator; Hydrosun Medizinaltechnik, Müllheim, Germany)
  Arms: wIRA irradiation
Other: visible light only — visible light application at a distance of 27cm from the skin surface with for 20 min.
  Other Names: Standard light bulb with visible normal conventional light.
  Arms: visible light only

SUMMARY:
The purpose of this study is to dermine whether local-water filtered infrared-A (wIRA) irradiation can reduce postoperative wound infection. wIRA irradiation is applied 20min directly preoperatively, before patients underwent abdominal surgery. The wIRA is a harmless light source, that has been described before. We test the impact and clinical outcome of patients undergoing a one-time preoperative wIRA irradiation on postoperative wound healing.

DETAILED DESCRIPTION:
Wound healing is a complex pathophysiological process that is related to pain, discomfort and immobility of patients and when not well controlled may lead to devastating and morbidity related wound infections. Furthermore, prolonged hospital stay, increased pain and consecutive increased drug consumption is often associated with postoperative wound infections. Although the average costs of wound infections are difficult to assess, there is no doubt that a prophylactic tool in controlling postoperative wound healing would have tremendous potential. Recent studies indicate that the application of different forms of thermal energy to the skin surface decreases postoperative wound infections significantly. It is known that high-normal arterial oxygen tension levels have decreased surgical wound infection from 11% to 5%. The application of water-filtered infrared A (wIRA) irradiation has been successfully applied in patients with ulcus cruris and superficial skin-tumors to alleviate pain and regulation of the body temperature in neonatology. The simple preoperative whole body warming for 30 min before surgery resulted in a statistically reduced occurrence of postoperative wound infections. A more recent study showed the beneficial effects of postoperative wIRA application on wound healing. The effects of wIRA leading to this success in therapy can be explained by thermal and non-thermal effects. A major advantage of the wIRA vs. the application of simple warming blankets lies upon the effective penetration of the wIRA applied energy within the deep subcutaneous tissue at depths of 2-3 cm. Further effects of the applied energy lead to vasodilation of capillaries with consecutive effective conduction of energetic blood flow into deeper tissue layers. Non-thermal effects of the wIRA application consist of direct stimulation and active immunomodulation by specialized immune cells. Furthermore, wIRA can induce protective proteins, e.g. ferritin in the skin and potentially influences common cross-talks within cells and extracellular matrices. These effects display regulatory roles in wound repair processes that may also be responsible for positive cosmetic results. More important for the clinical assessment of wound healing in the early phase of hospitalization is the effect of wIRA to significantly reduce postoperative pain. Surgery and postoperative pain evoke stress related effects that are induced by profound neuroendocrine changes in cytokine activity and related processes. Increased blood flow, due to vasodilation, helps to strongly eliminate accumulated pain mediators, lactic acid and potential bacterial toxins. The metabolism is induced and mediates also non-thermal effects such as attraction of immune cells and potential effects on nociceptors. These direct effects of wIRA can be easily followed when postoperative irradiation is performed. The problem of developing wound infections may rely within the first hours after and already during the operation, when the wound gets "preconditioned" with potential mediators or bacteria that may lead to postoperative encountered wound infections. A recent study indicated that immediate postoperative warming for 2 hours after hernia surgery may provide comparable benefits to seven days of warming. According to the idea of preventing deleterious preconditions in the process of wound healing, we tested here, the one time preoperative application of wIRA and its impact on postoperative wound healing and related clinical questions. Comparable to preoperative antibiotic single shot treatment we relied on the expansive impact of preoperative wIRA application.

The prospective randomized controlled clinical trial is designed to study the effects of single time preoperative wIRA irradiation on the postoperative outcome of wound infections after visceral surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing aseptic surgery with a median or transverse laparotomy
* informed consent
* Patients age between 30 and 80 years

Exclusion Criteria:

* pregnancy
* laparoscopic surgery
* operation time more than 6 hours
* signs of infection (local or systemic)
* MRSA positive patients
* myocardial infarction within 6 wks prior to surgery
* radio- or chemotherapy within 4 wks prior to surgery
* body temperature above 38°C for the last 5 days prior to surgery
* cachexia
* leucocytopenia
* liver cirrhosis Child B or C

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Postoperative wound infection rate | day 2 to 8 and day 30
  The rate of wound infection was assessed from day 2 to 8 and day 30 post surgery.
  The wound infection rate was assessed by a visual analogue scale (VAS) Group A: irradiated with local water-filtered infrared A (wIRA) irradiation Group B: irriadiate with conventional visible light

SECONDARY OUTCOMES:
Wound pain postoperative | day 2 to 8 and after 30 days
  Wound pain was assessed at day 2 to 8 (on a daily basis) and after day 30 post surgery, comparing patients from Group A (wIRA) and group B (only conventional light) application.
Wound healing postoperative | day 2 to 8 and after 30 days
  Wound healing was assessed at day 2 - 8 (daily) and after 30 days with a visual analogue scale (VAS).
  The wound healing was assessed while comparing the results from group A (wIRA) and group B (conventional light).

CONTACTS AND LOCATIONS:
Overall Officials: Beat M Künzli, MD, Study Director — Klinikum rechts der Isar, Technische Universität München, Munich, Germany
Locations (1):
- Klinikum rechts der Isar der Technischen Universität, Munich, Bavaria, Germany

REFERENCES:
- [Background] Hartel M, Hoffmann G, Wente MN, Martignoni ME, Buchler MW, Friess H. Randomized clinical trial of the influence of local water-filtered infrared A irradiation on wound healing after abdominal surgery. Br J Surg. 2006 Aug;93(8):952-60. doi: 10.1002/bjs.5429. PMID 16845694
- [Derived] Kunzli BM, Liebl F, Nuhn P, Schuster T, Friess H, Hartel M. Impact of preoperative local water-filtered infrared A irradiation on postoperative wound healing: a randomized patient- and observer-blinded controlled clinical trial. Ann Surg. 2013 Dec;258(6):887-94. doi: 10.1097/SLA.0000000000000235. PMID 24169161